CLINICAL TRIAL: NCT04196738
Title: Comparison of Volume Assist Control, Dual Mode and Airway Pressure Release Ventilation: A Physiological Study
Brief Title: Comparison of Volume Assist Control, Dual Mode and Airway Pressure Release Ventilation.
Acronym: COMIX-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 49RC19_0195
Record Dates: First submitted 2019-11-12; First posted 2019-12-12 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: ARDS

STUDY DESIGN:
Intervention Model Description: patients exposed to 3 ventilatory mode in 2 different possible orders
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Mode first (Experimental): Four consecutive steps (45 min per step) in the following order: APRV (A), Dual Mode (B) , APRV (A) and VAC (C). (ABAC)
  Interventions: Other: ventilation strategy
- VAC fist (Experimental): Four consecutive steps (45 min per step) in the following order: APRV (A), VAC (C) , APRV (A) and Dual Mode (B). (ACAB)
  Interventions: Other: ventilation strategy

INTERVENTIONS:
Other: ventilation strategy — Patients are ventilated in randomised order with three different ventilation strategies: volume assist control (constant flow), Dual Mode or Airway Pressure Released Ventilation

SUMMARY:
The aim of the COMIX-R study is to assess the short term physiological effects of 3 ventilation strategies for adult patients with ARDS admitted to intensive care unit

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Invasive mechanical ventilation on tracheal probe
* Acute respiratory distress syndrome, as defined by Berlin conference consensus, during hospitalization in intensive care,
* Recovery phase of acute respiratory distress syndrome: spontaneous ventilation representing from 20 to 30% of ventilation in APRV mode.
* No severe acidosis (pH> 7.30)
* Patient affiliated to or beneficiary of a health care plan
* Express consent of the patient or his/her SDM

Exclusion Criteria:

* Pneumothorax
* Contraindication to the insertion of a nasogastric tube with an esophageal balloon
* Contraindication to the use of Electrical impedance tomography (pacemaker)
* Pregnancy, lactating or parturient woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
change of PaO2 (mmHg) | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  Arterial partial pressure of dioxygen Of note: As it is a physiological study, all the primary and secondary outcomes will be analyzed with the same importance.

SECONDARY OUTCOMES:
-Respiratory rate variability | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  variability of rate (per minute)
-expiratory and inspiratory transpulmonary pressure | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  calculated with the esophageal pressure (cm H20)
-ventilation distribution in the lungs | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  Electrical impedance tomography (EIT) assess distribution of tidal volume and of end-expiratory lung volume (EELV) (delta Z, IU)
-other arterial parameters of hematosis | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  pH, PaO2, PaCo2 (mmHg)
-Work of breathing (WOB) | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  calculated with esophageal pressure (Kg/m)
-Pressure time product (PTP) | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  -Pressure time product (PTP) calculated with esophageal pressure (cmH2O.s.min-1)
-P0.1 | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  pressure measured during the first 100 ms after an occlusion (cm H20)
-PEEPi | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  intrinsic positive end-expiratory pressure (cm H20)
MAP | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  mean arterial pressure
HR | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  heart rate (beats per minute)
-Respiratory comfort | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  visual analogic scale
-Patient-ventilator asynchronies | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  numbers of asynchronies analyzed on screen
-Tidal volume variability | 15 minutes, 1 hour, 1hour and 45 minutes, 2 hour and 30 minutes
  variability of Tidal volume (mL)

CONTACTS AND LOCATIONS:
Overall Officials: Francois BELONCLE, CCU-AH, Principal Investigator — Angers teatching hospital
Locations (1):
- University hospital, Angers, France